CLINICAL TRIAL: NCT04665518
Title: The Effect of Acupressure on Acute Pain, Stress and Satisfaction During Venipuncture : Single-blind, Randomised Controlled Study
Brief Title: The Effect of Acupressure on Acute Pain, Stress and Satisfaction During Venipuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Prof. Dr., Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IZU01
Record Dates: First submitted 2020-11-23; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Pain, Acute; Satisfaction, Patient; Stress
Keywords: Acupressure; acute pain; stress; satisfaction; nursing; nonpharmacological methods
MeSH Terms: conditions — Acute Pain; Patient Satisfaction; Personal Satisfaction | interventions — Acupressure; Phlebotomy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): The following applications will be made 10 minutes before the patients in the acupressure group. Hands are washed before applying acupressure. Before acupressure is applied, the patient is allowed to sit in a comfortable position on the sofa in the single blood collection room. Before starting the acupressure application, the arm is rubbed from fingertips to the elbow to relax, and press the acupressure points (Large Intestine Meridian 4th Point [LI 4], Large Intestine Meridian 11th Point [LI 11], and Heart Meridian 7th Point [HT 7]). application is carried out. 2 minutes to each acupressure point. pressure (3 to 5 kg of pressure) is applied. Only one acupressure session is given to each patient, and each acupressure session lasts 10 minutes. Venipuncture is applied to all patients by the same nurse in the same room. Venipuncture is performed from the left arm of all patients using a vacuum tube and a needle tip of 0.8 * 38 mm (21G x 1½, green).
  Interventions: Other: Acupressure
- Control group (No Intervention): Venipuncture is applied to all patients by the same nurse in the same room. Venipuncture is performed from the left arm of all patients using a vacuum tube and a needle tip of 0.8 * 38 mm (21G x 1½, green).

INTERVENTIONS:
Other: Acupressure — Acupressure will be applied to the patients in the acupressure group for 10 min before the venipuncture procedure. Venipuncuture is applied to all patients by the same nurse in the same room. Venipuncture is performed from the left arm of all patients using a vacuum tube and a needle tip of 0.8 * 38 mm (21G x 1½, green).
  Other Names: Venipuncture
  Arms: Acupressure group

SUMMARY:
Acupressure, which is a type of nonpharmacological practice. Acupressure is a practice that provides energy flow by applying pressure to the special points of the meridians that innately carry energy in the body with stimulation bands, hands, and fingers. Acupressure is also known as acupuncture without needles. Because no needles are used in acupressure, acupressure is an easy, safe, effective, and economical method to learn and apply. There is no study to determine the effect of acupressure on acute pain, patient satisfaction and stress, which is applied to adult patients during the venipuncture procedure. In this context, the study was planned to be conducted in a randomized controlled trial to evaluate the effect of acupressure on acute pain, stress level and satisfaction during venpuncture in adult patients.Patient Evaluation Form, Visual Analogue Scale (VAS), Visual Patient Satisfaction Scale and State Anxiety Inventory will be used in the study. The scales will be used before and after venpuncture. Acupressure will be applied to the adults in the acupressure group for 10 min before the venipuncture procedure. Pain, heart rate, and oxygen saturation levels of the adults in the acupressure and control groups will be evaluated both before and after the venipuncture procedure.

DETAILED DESCRIPTION:
Patients will be assigned to acupressure and control groups according to the randomization list prepared earlier by the investigators.

First of all, all patients will be informed about the procedure and their informed consent will be obtained. Patients in the acupuncture and control groups will be evaluated with the patient evaluation form, VAS and State Anxiety Inventory 15 minutes before venipuncture. Demographic information of each patient will be recorded by the investigator. The pain level, satisfaction level and anxiety levels of the patients will be recorded before the venipuncture procedure. The following applications will be made 10 minutes before the patients in the acupressure group. Hands are washed before applying acupressure. Before applying acupressure, the patient is allowed to sit in a comfortable position on the sofa in the single venipuncture room. Before starting the acupressure application, the arm is rubbed from fingertips to the elbow to relax, and press the acupressure points (Large Intestine Meridian 4th Point [LI 4], Large Intestine Meridian 11th Point [LI 11], and Heart Meridian 7th Point [HT 7]). application is carried out. 2 minutes to each acupressure point. pressure (3 to 5 kg of pressure) is applied. Only one acupressure session is performed for each patient, and each acupressure session will last 10 minutes (WHO, 2008). Acupressure application is applied before venipuncture. Venipuncturen is performed immediately after the acupressure session. While performing the acupuncture procedure and venipuncture, other patients participating in the study will not see each other during the application phase. Venipuncture will be applied to all patients by the same nurse in the same room. Venipuncture will be performed on the left arm of all patients with a vacuum tube using a 0.8 * 38 mm (21G x 1½, green) needle tip. Immediately after the venipuncture, the pain and satisfaction assessment of the patients during the procedure will be made with the VAS (Pain and Satisfaction) and State Anxiety Inventory. The pain level, satisfaction level and anxiety levels of the patients will be recorded before the venipuncture procedure. All of the measurement results were obtained by another researcher blinded to group allocation. All procedures will take approximately 20-25 minutes for each participant.

ELIGIBILITY:
Inclusion Criteria:

* volunteer
* have not had venipuncture in the last 1 week

Exclusion Criteria:

* Patients with psychological and communication problems will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Before Assessment | 15 minutes before venipuncture
  Patients in the acupuncture and control groups will be evaluated with the sociodemographic form 15 minutes before venipuncture.
  It was prepared by the researchers by investigating the related literature and studies. In the form, there are 5 questions including some socio-demographic characteristics of the individuals (age, gender, marital status, educational background, BMI).
Before Assessment | 15 minutes before venipuncture
  Patients in the acupuncture and control groups will be evaluated with the Visual Anolog Scale for pain assessment 15 minutes before venipuncture. The scale is composed of a 10-cm horizontal or vertical line that starts with "No Pain" and ends with "Worst Pain". The use of Visual Anolog Scale should be explained to the patient very well. The patient is asked to mark his/her pain level on an appropriate point on this line. The distance between the beginning point of "no pain" and this point was measured and recorded as "10". Values range between 0 and 10 and the pain levels of the patients are evaluated over 10 points as 0 = no pain, 10 = worst pain.
Before Assessment | 15 minutes before venipuncture
  The satisfaction assessment of the patients during the procedure will be made with the Visual Analog Patient Satisfaction Scale form 15 minutes before venipuncture.
  Visual analog patient satisfaction scale is combined with the features of the well-known Visual Analog Patient Satisfaction Scale . It is composed of a 10 cm horizontal line without numbers. The expression of "I am very dissatisfied" is on one end of the line and the expression of "I am very satisfied" is on the other end. The patient should determine his/her satisfaction level by synthesizing all components affecting him/herself about the medical care given and find the point on line corresponding to his/her condition.
Before Assessment | 15 minutes before venipuncture
  Patients in the acupuncture and control groups will be evaluated with the State Anxiety Inventory to assess anxiety 15 minutes before venipuncture. The State Anxiety Scale consists of 20 questions about emotions, thoughts, and behaviors which are related to anxiety. The choices on this scale range from 1 (no anxiety) to 4 (extreme anxiety). Possible scores on the Scale range from 0 to 19 points (interpreted as meaning no state anxiety), 20 to 39 points (mild), 40 to 59 points (moderate), 60 to 79 points (severe), and 80 points and azbove (very severe state anxiety).
After Assessment | 5 minutes after venipuncture
  The pain assessment of the patients during the procedure will be made with the Visual Analog Scale within 5 minutes after the venipuncture.
  The scale is composed of a 10 cm horizontal or vertical line that starts with "No Pain" and ends with "Worst Pain". The use of Visual Anolog Scale should be explained to the patient very well. The patient is asked to mark his/her pain level on an appropriate point on this line. The distance between the beginning point of "no pain" and this point was measured and recorded as "10". Values range between 0 and 10 and the pain levels of the patients are evaluated over 10 points as 0 = no pain, 10 = worst pain.
After Assessment | 5 minutes after venipuncture
  The satisfaction assessment of the patients during the procedure will be made with the Visual Analog Patient Satisfaction Scale within 5 minutes after the venipuncture.
  Visual Analog Patient Satisfaction scale is combined with the features of the well-known Visual Analog Patient Satisfaction Scale . It is composed of a 10 cm horizontal line without numbers. The expression of "I am very dissatisfied" is on one end of the line and the expression of "I am very satisfied" is on the other end. The patient should determine his/her satisfaction level by synthesizing all components affecting him/herself about the medical care given and find the point on line corresponding to his/her condition.
After Assessment | 5 minutes after venipuncture
  Patients in the acupuncture and control groups will be evaluated with the State Anxiety Inventory to assess anxiety within 5 minutes after the venipuncture.
  The State Anxiety Scale consists of 20 questions about emotions, thoughts, and behaviors which are related to anxiety. The choices on this scale range from 1 (no anxiety) to 4 (extreme anxiety). Possible scores on the Scale range from 0 to 19 points (interpreted as meaning no state anxiety), 20 to 39 points (mild), 40 to 59 points (moderate), 60 to 79 points (severe), and 80 points and azbove (very severe state anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yıldırım, Principal Investigator
Locations (1):
- Dilek Yıldırım, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koc Ozkan T, Balci S. The Effect of Acupressure on Acute Pain During Venipuncture in Children: Implications for Evidence-Based Practice. Worldviews Evid Based Nurs. 2020 Jun;17(3):221-228. doi: 10.1111/wvn.12437. Epub 2020 Apr 22. PMID 32320139